CLINICAL TRIAL: NCT03094208
Title: Investigation of the Effects of Dual Task Balance Training In Indıvıduals With Above Knee Amputation
Brief Title: The Effects of Dual Task Balance Training In Individuals With Above Knee Amputation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Senem Demirdel, Hacettepe University, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO16/641-16
Record Dates: First submitted 2017-03-15; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Amputation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): muscle strengthening, weight transfer, dual task balance exercises, dual task gait exercises.
  Interventions: Other: dual task balance training
- control group (Active Comparator): muscle strengthening, weight transfer, balance exercises, gait exercises.
  Interventions: Other: traditional balance training

INTERVENTIONS:
Other: dual task balance training — balance exercises with cognitive and motor dual tasks
  Other Names: Study group will also receive dual task balance training
  Arms: study group
Other: traditional balance training — balance exercises
  Arms: control group

SUMMARY:
The people with transfemoral amputation who use mechanical prosthesis will be include to this study. All participants will be assessed and then they will be randomly assigned to two groups. both groups will receive traditional balance trainnig. Study group will also receive dual task balance training. Training will take 4 weeks, 3 days a week. After the training program, both groups will be assessed again and the results will compare.

DETAILED DESCRIPTION:
The people who have transfemoral amputation may have poor balance and gait. Many people with lower limb loss report the need to concentration on gait. People with lower limb loss may need to use cognitive resources to monitor and control movements of the prosthetic limb. The need to concentrate on walking may be greater for those with transfemoral amputation. For examine the use of cognitive resources, dual task paradigm may use. Dual task rehabilitative training used in many patients like stroke, Multipl sclerosis osteoporosis. But there is no study about dual task training on amputation. The purpose of this randomized controlled study is to investigate the effects of dual-task balance training on balance and gait of patients with transfemoral amputation as compared with single-task balance training. We hypothesized that dual-task balance training would improve the balance and gait, it would be more effective than single-task balance training.

ELIGIBILITY:
Inclusion Criteria:

* Peoples with transfemoral amputations
* people who use their mechanical prosthetics at least 1 year
* People who can walk withoud aids

Exclusion Criteria:

* People who have the other health conditions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-16 (Estimated); Primary Completion 2018-06-15 (Estimated); Study Completion 2018-08-15 (Estimated)

PRIMARY OUTCOMES:
gait speed | 1 minute
  10 meter walk test

SECONDARY OUTCOMES:
gait analysis | 1 minute
  gait analysis with footprint method
cognition | 5 minutes
  Montreal Cognitive Assessment
depression | 3 minutes
  Beck Depression invertory
balance | 2 minutes
  one leg stance test
balance | 1 minute
  four square step test
functional mobility | 1 minute
  timed up and go test

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Erbahçeci, Prof, Principal Investigator — Hacettepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morgan SJ, Hafner BJ, Kelly VE. The effects of a concurrent task on walking in persons with transfemoral amputation compared to persons without limb loss. Prosthet Orthot Int. 2016 Aug;40(4):490-6. doi: 10.1177/0309364615596066. Epub 2015 Jul 24. PMID 26209423
- [Background] Kim GY, Han MR, Lee HG. Effect of Dual-task Rehabilitative Training on Cognitive and Motor Function of Stroke Patients. J Phys Ther Sci. 2014 Jan;26(1):1-6. doi: 10.1589/jpts.26.1. Epub 2014 Feb 6. PMID 24567664
- [Background] Monjezi S, Negahban H, Tajali S, Yadollahpour N, Majdinasab N. Effects of dual-task balance training on postural performance in patients with Multiple Sclerosis: a double-blind, randomized controlled pilot trial. Clin Rehabil. 2017 Feb;31(2):234-241. doi: 10.1177/0269215516639735. Epub 2016 Jul 10. PMID 27006419
- [Derived] Demirdel S, Erbahceci F. Investigation of the Effects of Dual-Task Balance Training on Gait and Balance in Transfemoral Amputees: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2020 Oct;101(10):1675-1682. doi: 10.1016/j.apmr.2020.06.009. Epub 2020 Jul 10. PMID 32653580